CLINICAL TRIAL: NCT06582329
Title: Effect of Alpha-1 Antitrypsin Supplementation on Alcohol-Associated Hepatitis - A Prospective Pilot Study
Brief Title: Effect of Alpha-1 Antitrypsin Supplementation on Alcohol-Associated Hepatitis
Acronym: EARTH
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EARTH-2024
Record Dates: First submitted 2024-07-31; First posted 2024-09-03 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-08

CONDITIONS: Alcohol-Associated Hepatitis
MeSH Terms: interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Intervention Model Description: Therapeutic exploratory trial:
  the trial is designed as a prospective, single center, open label, randomized controlled pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard of care (No Intervention): Standard of care Prednisolon 40mg will be administered over 4 weeks
- Standard of care + Alpha 1 Antitrypsin (Experimental): In the experimental arm the participants will receive Prolastin 120 mg/kg bodyweight and Prednisolon 40 mg over a time period of 4 weeks
  Interventions: Drug: Alfa1 Antitrypsin

INTERVENTIONS:
Drug: Alfa1 Antitrypsin — Participants will be treated intravenously with A1AT 120 mg/kg bodyweight once a week for 4 weeks (4 total infusions).
  Arms: Standard of care + Alpha 1 Antitrypsin

SUMMARY:
The trial is designed as a prospective, single center, open label, randomized controlled pilot study evaluating the effect of A1AT (Alpha 1 Antitrypsin) on inflammation in patients with severe AAH (alcohol-associated hepatitis).

The objective is to evaluate the safety and the effect of intravenous A1AT on the systemic inflammation in patients with severe AAH. The objectives also include the assessment of A1AT on clinical outcomes including the incidence of adverse events (AEs) and serious adverse events (SAEs) and the cytokine.

DETAILED DESCRIPTION:
About 5-7 % of patients with alcohol-associated chronic liver disease transform into acute on chronic liver disease (ACLF) per year. In patients with underlying alcohol-associated liver disease (ALD) and active drinking, a sudden onset of jaundice, malaise, decompensated liver disease and coagulopathy i.e. alcohol-associated hepatitis (AAH) might develop. In its severe form, AAH is associated with development of ACLF and bacterial infections and this disease exhibits a high short-term mortality of 20 to 50% within 3 months. Treatment options are limited currently, for instance, the use of corticosteroids.

Alpha-1 Antitrypsin (A1AT) acts as an anti-inflammatory protein by inhibiting the generation of pro-inflammatory cytokines. The investigators recently showed protective effects of A1AT in a pre-clinical experimental model of ALD, resulting in decreased levels of pro-inflammatory cytokines, less steatosis and hepatic injury. The investigators also have recently found that cirrhotic patients with A1AT concentrations less than 120 mg/dL had a significantly increased risk for death/liver transplantation in a cohort of 130 patients with ALD cirrhosis. This finding was not only significant, but also independent of the MELD-Na score, indicating that in ALD A1AT is not only a marker of reduced hepatic synthetic function. Further, significantly higher ferritin and lower transferrin in the cohort of patients with low A1AT also indicate more severe inflammation. An interventional analysis in an established mouse model of ALD showed that A1AT supplementation mitigated inflammation and histological changes further indicating that low AAT (Alpha 1 Antitrypsin) is a driver and not the consequence of tissue damage in ALD. These data support the use of A1AT in humans with severe AAH.

As a pilot trial the study also aims to establish important preliminary data for future studies and design of larger trials aimed at formal evaluation of the effect of A1AT on clinical endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient ≥18 years of age at time of consent.
2. Severe AAH (Maddrey's discriminant function score ≥ 32) at screening.
3. No ACLF or ACLF Grade 1 at screening.
4. Daily average intake of >80 g (men)/>60 g (women) ethanol during the past 3 months (patient reported).
5. Understands and agrees to comply with the study procedures and provides written informed consent as documented by signature.
6. Outpatient or hospitalized patient not being on the Intensive Care Unit (ICU) at screening.

   Inclusion criterion 7 only applies to women of childbearing potential (WOCBP)
7. Negative urine pregnancy test, not breastfeeding & agreement to use highly-effective means of contraception during the study. Allowed are sexual abstinence, vasectomized partners (˃3 months previously-vasectomy has to be confirmed by two negative semen analyses) or the consistent and correct use of an approved contraceptive method in accordance with the product label, for example: Barrier method (such as condoms, diaphragm, or cervical cap) used in conjunction with spermicide; intrauterine device; prescription hormonal contraceptive taken or administered via oral (pill), transdermal (patch), subdermal, or intramuscular (IM) route Inclusion criterion 8 only applies to male patients
8. Male patients who are sexually active with female partners of childbearing potential must agree to use a condom with spermicide and to use one other approved method of highly effective contraception from the time of investigational product administration for at least 90 days after the dose of investigational product and must refrain from sperm donation from Screening through at least 90 days following the last dose of investigational product.
9. Ability to speak and read German to a level which allows fully comprehending the meaning of everything that is said and written.

Exclusion Criteria:

1. Uncontrolled Diabetes Mellitus type 1 or 2 (defined by HbA1c > 10%).
2. Corticosteroid use contraindicated.
3. Viral hepatitis, autoimmune hepatitis, HIV infection, Wilson disease, hemochromatosis, toxic liver injury, Primary Biliary Cholangitis (PBC), Primary Sclerosing Cholangitis (PSC).
4. Participation in another interventional clinical study within 6 months prior to screening and/or during trial participation.
5. Presence of any active malignancy (other than non-melanoma skin cancer) which required treatment within the past 12 months.
6. Chronic kidney disease receiving dialysis.
7. Do Not Attempt Resuscitation (DNAR) order in place.
8. IgA deficiency (IgA level <7mg/dL) or known intolerance to A1AT.
9. History of liver transplantation or currently listed for liver transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Serum concentration of IL-6 (interleukin-6) assessed at Visit 2 (Day 8+/-1) in the intervention (A1AT in combination with standard-of-care) and control group (standard-of-care). | at visit 2
  The effect on the serum IL-6 concentration assessed after 1 week will be assessed at Visit 2 (Day 8+/-1) in the intervention (A1AT in combination with standard-of-care) and control group (standard-of-care).

SECONDARY OUTCOMES:
Serum A1AT concentration assessed at visit 5 (Day 29+/-3) | at visit 5 (Day 29+/-3)
Incidence of Adverse Events (AEs) from the baseline visit (Day 1) to end of study visit (Day 90+/-7) | up to 3 months
Incidence of Serious Adverse Events (SAEs) from the baseline visit (Day 1) through to end of study visit (Day 90+/-7) | up to 3 months
Chronic Liver Disease Questionnaire (CLDQ) overall and subscale scores. | up to 3 months
  The response of CLDQ results in 1 to 7 scales, ranging from "all the time" to "none of the time". Higher scores indicate the minimum frequency of symptoms and therefore a better HRQL
CLDQ-D overall and subscale scores | up to 3 months
  The response of CLDQ results in 1 to 7 scales, ranging from "all the time" to "none of the time". Higher scores indicate the minimum frequency of symptoms and therefore a better HRQL.

OTHER OUTCOMES:
Model for end-stage liver disease (MELD) | up to 3 months
  The Model for End-Stage Liver Disease (MELD) is a numerical scale, ranging from 6 (you are less sick) to 40 (you are gravely sick), used for liver transplant candidates
The MELD-sodium (MELD-Na) | up to 3 months
  MELD-Na Score adds sodium to the MELD model for liver cirrhosis. The Model for End-Stage Liver Disease (MELD) is a numerical scale, ranging from 6 (you are less sick) to 40 (you are gravely sick), used for liver transplant
Child-Pugh-Turcotte | up to 3 months
  The score employs five clinical measures of liver disease. Each measure is scored 1-3, with 3 indicating most severe derangement. Chronic liver disease is classified into Child-Pugh class A to C, employing the added score from above. 5-6 points class A, 79 points class B, 10-15 points class C. Class A with the best outcome, class C with the most severe.
CLIF (Chronic Liver Failure)-C-AD (acute decompensation) | up to 3 months
  The CLIF-C acute decompensation (AD) score is used to predict prognosis of patients with acute decompensation of cirrhosis who do not have acute-on-chronic liver failure (ACLF).
CLIF-C-OF (organ function) | up to 3 months
  Each organ system is scored on a scale to generate the overall CLIF-C OF score, ranging from 0 to 18. A higher CLIF-C OF score translates into a higher ACLF grade.
CLIF-SOFA (Sequential Organ Failure Assessment) score | up to 3 months
  The CLIF-SOFA score is calculated on a scale from 0 to 4, whereas 4 means the worst outcome
Maddrey's discriminant function | up to 3 months
  Prospective studies have shown that it is useful in predicting short term prognosis, especially mortality within 30 days. A value more than 32 implies poor outcome
Time to hospital discharge | up to 3 months
Time to re-hospitalization | up to 3 months
Time to ICU admission | up to 3 months
Liver-specific survival and transplant-free survival at End of Study Visit | up to 3 months
Serum concentrations of IL-6 | up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck, Innsbruck, Austria